CLINICAL TRIAL: NCT00763386
Title: Prospective Randomized Multicenter Study of NexGen LPS-Flex Knee
Brief Title: A Study to Compare the NexGen LPS and LPS-Flex Knee Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00-500
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: Total Knee Arthroplasty; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Study arm will consist of patients that are treated with the NexGen LPS-Flex Fixed Bearing Knee.
  Interventions: Device: NexGen LPS-Flex Fixed Bearing Knee
- 2 (Active Comparator): Study arm will consist of patients that are treated with the NexGen Legacy Posterior Stabilized Knee.
  Interventions: Device: NexGen Legacy Posterior Stabilized Knee

INTERVENTIONS:
Device: NexGen LPS-Flex Fixed Bearing Knee — NexGen LPS-Flex Fixed Bearing femoral component
  Other Names: LPS-Flex Knee
  Arms: 1
Device: NexGen Legacy Posterior Stabilized Knee — NexGen Legacy Posterior Stabilized femoral component
  Other Names: LPS Knee
  Arms: 2

SUMMARY:
The purpose of this study is to test for significant differences in functional outcomes obtained by using a NexGen LPS versus a NexGen LPS-Flex knee implant. Specifically, it is predicted that an increase in postoperative range of motion will be experienced by patients treated with the NexGen LPS-Flex knee implant.

DETAILED DESCRIPTION:
This study will compare the clinical results of the NexGen LPS femoral component with the higher flexion potential of the NexGen LPS-Flex femoral component in all patients with degenerative joint disease that require total knee arthroplasty. The primary variable of interest is postoperative range of motion achieved with the two devices, which are implanted with slightly different surgical techniques in patients who may also be subjected to different rehabilitation programs depending on the device they are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Age, 21-80 years
* Sex, Males and females will be included
* BMI less than or equal to 39 and calf-thigh less than or equal to 90 degrees
* Stable health, the patient would be able to undergo surgery and participate in the follow-up program based on physical examination and medical history.
* Patient is willing and able to cooperate in follow-up therapy.
* Patient exhibits preoperative radiographic evidence of joint degeneration consistent with TKA that cannot be treated in non-operative fashion.
* Patient has stable and functional collateral ligaments.
* Patient has potential to perform higher than average range of motion activities.
* Operative side range of motion flexion greater than or equal to 90 degrees.
* Severe knee pain and disability due to degenerative joint disease.
* Patient or patient's legal representative has signed the Informed Consent form.

Exclusion Criteria:

* Previous history of infection in the affected joint.
* Previously failed knee endoprosthesis of any kind.
* Charcot joint disease or other severe neurosensory deficits.
* Previous patellectomy.
* Patient is skeletally immature.
* Grossly insufficient femoral or tibial bone stock.
* Patient is pregnant.
* Varus or valgus deformity greater than 20 degrees.
* Fixed flexion deformity greater than 15 degrees.
* Previous high tibial osteotomy.
* Previous femoral osteotomy.
* Patient is a poor compliance risk - currently treated for ethanol or drug abuse, physical or mental handicap, etc.
* Loss of musculature or absence of musculoligamentous supporting structures required for adequate soft tissue balance.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2001-06; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - VA Medical Center, Decatur, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Joint Replacement Surgeons of Indiana, Indianapolis, Indiana
  - The Center for Hip and Knee Surgery, Mooresville, Indiana
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - VSAS Orthopaedics, Allentown, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Piedmont Orthopaedic Associates, Greenville, South Carolina
  - Orthopaedic Specialists of Spartanburg, Spartanburg, South Carolina
  - Vanderbilt Orthopaedic Institute, Nashville, Tennessee
  - Rebecca Sealy Hospital, Galveston, Texas
  - The Rectors and Visitors of the University of Virginia, Charlottesville, Virginia
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between June 2001 and December 2007 at a total of 12 sites throughout the US/Canada
Groups:
- LPS Flex Fixed Bearing Knee: Study arm will consist of patients that are treated with the NexGen LPS-Flex Fixed Bearing Knee.
- LPS Standard Knee: Study arm will consist of patients that are treated with the NexGen Legacy Posterior Stabilized Knee.
Period: Overall Study
Arm/Group | LPS Flex Fixed Bearing Knee | LPS Standard Knee
Started | 164 | 167
Completed | 116 | 127
Not Completed | 48 | 40
Not completed — Adverse Event | 43 | 33
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — CRF missing | 0 | 1
Not completed — Study Prosthesis Removed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPS Flex Fixed Bearing Knee | LPS Standard Knee | Total
Number analyzed (Participants) | 164 | 167 | 331
Age Categorical [Number; unit: participants] — An LPS Standard patient's demographic CRF is missing and therefore, the total numbers for this category will be off by one.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 83 | 82 | 165
    >=65 years | 81 | 84 | 165
Age Continuous [Mean (Standard Deviation); unit: years] — An LPS Standard patient's demographic CRF is missing and therefore, the total numbers for this category will be off by one.
  years | 64.6 (8.1) | 64.9 (8.4) | 64.7 (8.3)
Gender [Number; unit: participants] — An LPS Standard patient's demographic CRF is missing and therefore, the total numbers for this category will be off by one.
  participants
    Female | 92 | 84 | 176
    Male | 72 | 82 | 154
Region of Enrollment [Number; unit: participants]
  United States | 133 | 138 | 271
  Canada | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Range of Motion (ROM)
Description: Postoperative ROM was calculated by taking the measurement of patient flexion minus the measurement of patients' extension.
Time Frame: 6 Weeks to 2 Years Post-op, based on on the intervals listed
Population: Analysis was determined by calculating the measurements of the enrolled cases who completed the stated visit interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | LPS Flex Fixed Bearing Knee | LPS Standard Knee
Number analyzed (Participants) | 164 | 167
degrees
  PostOp ROM @ 6 Weeks | 102.3 (17.1) | 106.8 (13.9)
  PostOp ROM @ 6 Months | 117.6 (11.3) | 118.2 (12.1)
  PostOp ROM @1 Year | 120.3 (10.7) | 121.7 (10.4)
  PostOp ROM @2 Year | 120.7 (10.7) | 121.2 (10.4)

2. Secondary Outcome: Return to Function (RtF) Via Knee Society Score (Modified)
Description: Scores were calculated from responses on a modified Knee Society Score by the enrolled subjects for the stated visit intervals.
  Grading for the Knee Society Score is based on a scale from 0-100 and results are established follows: 80-100 =Excellent; 70-79 = Good; 60-69 = Fair; and Below 60 = Poor.
Time Frame: 6 Weeks to 2 Years Post-op, based on on the intervals listed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LPS Flex Fixed Bearing Knee | LPS Standard Knee
Number analyzed (Participants) | 164 | 167
units on a scale
  PostOp KSSF @ 6 Week | 56.4 (21.7) | 58.5 (19.8)
  PostOp KSSF @ 6 Month | 79.2 (19.5) | 79.7 (20.0)
  PostOp KSSF @ 1 Year | 81.1 (21.9) | 81.7 (19.5)
  PostOp KSSF @ 2 Year | 84.3 (18.9) | 83.1 (18.9)

ADVERSE EVENTS:
Time Frame: Overall Study
Arm/Group | LPS Flex Fixed Bearing Knee | LPS Standard Knee
Serious Adverse Events (participants affected / at risk) | 13/164 | 19/167
Other Adverse Events (participants affected / at risk) | 27/164 | 23/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LPS Flex Fixed Bearing Knee (N=164) | LPS Standard Knee (N=167)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 2 (2)
Other Knee Related Complication (Musculoskeletal and Connective Tissue Disorders) (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
Stiff Knee Resulting in Manipulation (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Other General Complications (Musculoskeletal and Connective Tissue Disorder) (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (10)
Other General Complications (Neoplasms benign, malignant and unspecified) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Patellofemoral Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Quad Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other General Complication (Renal and Urinary Disorders) (Renal and urinary disorders) | 1 (1) | 1 (1)
Other General Complication (Surgical and Medical Procedures) (Surgical and medical procedures) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Other General Complication (Ear and Labyrthinth Disorders) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Other General Complication (Endocrine Disorders) (Endocrine disorders) | 0 (0) | 1 (1)
Patellar Implant Loosening (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other Knee Related Complication (Neoplasms benign, malignant and unspecified) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LPS Flex Fixed Bearing Knee (N=164) | LPS Standard Knee (N=167)
Other General Disorders (GI Disorder) (Gastrointestinal disorders) | 3 (6) | 0 (0)
Other General Complication (Musculoskeletal and Connective Tissue Disorder) (Musculoskeletal and connective tissue disorders) | 13 (27) | 12 (19)
Other Knee Related Complication (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Stiff Knee Resulting in Manipulations (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Other General Complication (Vascular Disorder) (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No